CLINICAL TRIAL: NCT04520997
Title: A Randomized, Evaluator-Blinded Study to Evaluate Facial Harmony and Subject Satisfaction Using Restylane Defyne in a Stepwise Treatment Approach
Brief Title: Restylane Defyne in a Stepwise Treatment Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05DF1910
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Lower Face Folds and Lines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Down-up (Experimental): Participants in this group received up to 2 mL Restylane Defyne on chin at baseline and up to 2 mL of Restylane Defyne per NLF at baseline and up to 2 mL per ML of Restylane Defyne at Week 3. An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator.
  Interventions: Device: Restylane Defyne
- Top-down (Experimental): Participants in this group received up to 2 mL Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at baseline and up to 2mL on chin Week 3. An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator.
  Interventions: Device: Restylane Defyne

INTERVENTIONS:
Device: Restylane Defyne — Up to 2 milliliters (ml) of Restylane Defyne per treatment site (chin and surrounding area) with maximum of total 4 ml at baseline, up to 2 ml of Restylane Defyne per NLF and ML at week 3 and optional up to 2 ml of Restylane Defyne per facial half for NLF and ML in combination with a total of 2 ml in the chin and surrounding area at week 6.
  Arms: Down-up
Device: Restylane Defyne — Up to 2 ml of Restylane Defyne per NLF and ML at baseline, up to 2 ml of Restylane Defyne per treatment site (chin and surrounding area) with maximum of total 4 ml at week 3 and optional touch-up of up to 2 ml per facial half for NLF and ML in combination with a total of 2 ml in the chin and surrounding area at week 6.
  Arms: Top-down

SUMMARY:
This was a 12-week study to evaluate the effectiveness and safety of Restylane Defyne when using two different injection approaches, stepwise down-up vs. top-down, when treating the lower face.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willed to comply with the requirements of the study and provided a signed written informed consent
* Subjects willed to undergo augmentation and correction therapy in the studied indications
* Adult males or non-pregnant, non-breastfeeding females and women of non-child bearing potential over the age of 21

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram-positive bacterial proteins
* Previous use of any permanent (non-biodegradable) treatment, lifting threads, permanent implants or autologous fat below the level of the horizontal line from the lower orbital rim
* Participation in any interventional clinical study within 30 days of screening

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Galderma Research Site, Birmingham, Alabama
  - Galderma Research Site, Chicago, Illinois
- Brazil (2):
  - Galderma Research Site, Belo Horizonte
  - Galderma Research Site, São Paulo
- Galderma Research Site, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 sites each in Brazil and Unites States,1 site in Italy from 07 Dec 2020 to 15 Sept 2021.
Groups:
- Down-up: Participants in this group received injections in the chin and surrounding area with up to 2 milliliters (mL) Restylane Defyne per treatment site with a maximum of 4 mL in total at Baseline and in the nasolabial folds (NLFs) and marionette lines (MLs) with up to 2 mL of Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at Week 3 (second injection). An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator at 6 weeks after second injection.
- Top-down: Participants in this group received injections in the NLFs and MLs with up to 2 mL of Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at Baseline and in the chin and surrounding area with up to 2 mL of Restylane Defyne per treatment site with a maximum of 4 mL in total at Week 3 (second injection). An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator at 6 weeks after second injection.
Period: Overall Study
Arm/Group | Down-up | Top-down
Started | 32 | 30
Treated (One participant randomized in Down-up but not treated.) | 31 | 29 (One participant was randomized to Top-down but was treated as Down-up. So, analysed according to the treatment received that is (i.e.), Down-up.)
Safety Population | 32 | 29
MITT (Modified Intention-to-treat) Population (One participant was withdrawn after first treatment in Down-up and therefore not included in MITT population.) | 31 | 29
Completed | 30 | 28
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: MITT population included all participants who were treated at both baseline and week 3.
Groups:
- Down-up: Participants in this group received injections in the chin and surrounding area with up to 2 mL Restylane Defyne per treatment site with a maximum of 4 mL in total at Baseline and in the NLFs and MLs with up to 2 mL of Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at Week 3 (second injection). An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator at 6 weeks after second injection.
- Total: Total of all reporting groups
Arm/Group | Down-up | Top-down | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.0) | 44.5 (11.4) | 44.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fitzpatrick Skin Types [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is a numerical classification scale for the color of skin from Type I to Type VI. Type I= always burns, never tans, Type II= usually burns, tans minimally (light colored but darker than fair), Type III= sometimes mild burn, tans uniformly (golden honey or olive), Type IV= burns minimally, always tan well (moderate brown), Type V= very rarely burns, tans very easily (dark brown), Type VI= never burns (deeply pigmented dark brown to darkest brown).
  Participants
    Type I | 0 | 2 | 2
    Type II | 11 | 7 | 18
    Type III | 10 | 14 | 24
    Type IV | 9 | 6 | 15
    Type V | 0 | 0 | 0
    Type VI | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Responders) With Aesthetic Improvement by the Treating Investigator Assessment Using Global Aesthetic Improvement Scale (GAIS) at Week 3
Description: Aesthetic improvement in chin and nasolabial fold/marionette line, and in combination was assessed on a 5-graded GAIS from "worse" to "very much improved" as follows; very much improved (optimal cosmetic result for the participant), much improved (marked improvement in appearance from the original condition, but not completely optimal for this participant), improved (obvious improvement in appearance from the original condition), no change (the appearance is essentially the same as the original condition), worse (the appearance is worse than the original condition). Responder was defined as a participant with a rating of at least improved as assessed by the treating investigator (assessed as very much improved, much improved or improved) compared to pre-treatment. Number of participants (responders) with aesthetic improvement based on treating investigator assessment using GAIS at Week 3 were reported.
Time Frame: At Week 3
Population: MITT population included all participants who were treated at both Baseline and Week 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Down-up | Top-down
Number analyzed (Participants) | 31 | 29
Participants
  Very Much Improved | 18 | 12
  Much Improved | 10 | 8
  Improved | 3 | 9

2. Primary Outcome: Percentage of Participants (Responders) With Aesthetic Improvement Based on Treating Investigator Assessment Using GAIS at Week 6
Description: Aesthetic improvement in chin and nasolabial fold/marionette line, and in combination was assessed on a 5-graded GAIS from "worse" to "very much improved" as follows; very much improved (optimal cosmetic result for the participant), much improved (marked improvement in appearance from the original condition, but not completely optimal for this participant), improved (obvious improvement in appearance from the original condition), no change (the appearance is essentially the same as the original condition), worse (the appearance is worse than the original condition). Responder was defined as a participant with a rating of at least improved as assessed by the Treating Investigator (assessed as very much improved, much improved or improved) compared to pre-treatment. Percentage of participants (responders) with aesthetic improvement based on treating investigator assessment using GAIS at Week 6 were reported.
Time Frame: At Week 6
Population: MITT population included all participants who were treated at both Baseline and Week 3. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Groups:
- Down-up: Participants in this group received injections in the chin and surrounding area with up to 2 mL Restylane Defyne per treatment site with a maximum of 4 mL in total at Baseline and in NLFs and MLs with up to 2 mL of Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at Week 3 (second injection). An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator at 6 weeks after second injection.
Arm/Group | Down-up | Top-down
Number analyzed (Participants) | 30 | 29
Percentage of participants
  Very Much Improved | 56.7 | 75.9
  Much Improved | 36.7 | 17.2
  Improved | 6.7 | 6.9

3. Primary Outcome: Percentage of Participants (Responders) With Aesthetic Improvement Based on Treating Investigator Assessment Using GAIS at Week 9
Description: Aesthetic improvement in chin and nasolabial fold/marionette line, and in combination was assessed on a 5-graded GAIS from "worse" to "very much improved" as follows; very much improved (optimal cosmetic result for the participant), much improved (marked improvement in appearance from the original condition, but not completely optimal for this participant), improved (obvious improvement in appearance from the original condition), no change (the appearance is essentially the same as the original condition), worse (the appearance is worse than the original condition). Responder was defined as a participant with a rating of at least improved as assessed by the Treating Investigator (assessed as very much improved, much improved or improved) compared to pre-treatment. Percentage of participants (responders) with aesthetic improvement based on treating investigator assessment using GAIS at Week 9 were reported.
Time Frame: At Week 9
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Down-up; Top-down: Participants in this group received injections in the NLFs and MLs with up to 2 mL of Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at Baseline and in the chin and surrounding area with up to 2 mL of Restylane Defyne per treatment site with a maximum of 4 mL in total at Week 3 (second injection). An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator at 6 weeks after second injection.
Arm/Group | Down-up | Top-down
Number analyzed (Participants) | 30 | 28
Percentage of participants
  Very Much Improved | 76.7 | 71.4
  Much Improved | 20.0 | 17.9
  Improved | 3.3 | 10.7

4. Secondary Outcome: Percentage of Participants With Naturalness of the Treatment Result as Assessed by Treating Investigator
Description: The treating investigator assessed the naturalness of the treatment result based on review of baseline photographs and live assessment on how much they agreed or disagreed to the statement as follows: "The treatment results were natural looking". The investigator's questionnaire for naturalness of the treatment result were categorized into "strongly agree, agree, neither agree or disagree, disagree and strongly disagree". The percentage of participants with naturalness of the treatment result as assessed by treating investigator were reported.
Time Frame: At Week 3, 6, and 9
Population: MITT population included all participants who were treated at both Baseline and Week 3. Here, "number analyzed" signifies participants who were evaluable for this outcome measure at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Down-up | Top-down
Number analyzed (Participants) | 31 | 29
Percentage of participants
  Naturalness at Week 3: Strongly agree | 90.3 | 89.7
  Naturalness at Week 3: Agree | 9.7 | 10.3
  Naturalness at Week 6: Strongly agree: number analyzed (Participants) | 30 | 29
  Naturalness at Week 6: Strongly agree | 90.0 | 89.7
  Naturalness at Week 6: Agree: number analyzed (Participants) | 30 | 29
  Naturalness at Week 6: Agree | 10.0 | 10.3
  Naturalness at Week 9: Strongly agree: number analyzed (Participants) | 30 | 28
  Naturalness at Week 9: Strongly agree | 73.3 | 89.3
  Naturalness at Week 9: Agree: number analyzed (Participants) | 30 | 28
  Naturalness at Week 9: Agree | 26.7 | 10.7

5. Secondary Outcome: Percentage of Participants Agreeing With Statements in a Satisfaction Questionnaire (SSQ)
Description: Participants completed 7 questions of subject satisfaction Questionnaire which are listed as follows: a) My first treatment improved my appearance, b) Compared to my first treatment, treating both areas in combination improved appearance, c) I am satisfied with the contour of my lower face after treatment, d) I am satisfied with the shape of my chin, e) I am satisfied with how well defined my chin looks, f) I feel more attractive after treatment, g) I feel comfortable being photographed. SSQ was balanced on 5-point scale assessing subject satisfaction with study treatment. Possible scores range was 1-Very Satisfied, 2-Satisfied, 3-Neither satisfied nor dissatisfied, 4-Dissatisfied, 5-Very Dissatisfied. Percentage of participants who strongly agreed or agreed to the SSQ were reported.
Time Frame: At Week 3, 6 and 9
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Groups:
- Down-up: Participants in this group received injections in the chin and surrounding area with up to 2 mL Restylane Defyne per treatment site with a maximum of 4 mL in total at Baseline and in the NLFs and marionette lines MLs with up to 2 mL of Restylane Defyne per NLF and up to 2 mL per ML of Restylane Defyne at Week 3 (second injection). An optional touch-up was administered to participants who had not achieved the optimal aesthetic improvement as agreed between participant and investigator at 6 weeks after second injection.
Arm/Group | Down-up | Top-down
Number analyzed (Participants) | 31 | 29
Percentage of participants
  My first treatment improved my appearance at Week 3 | 100 | 93.1
  My first treatment improved my appearance at Week 6: number analyzed (Participants) | 30 | 29
  My first treatment improved my appearance at Week 6 | 93.3 | 93.1
  My first treatment improved my appearance at Week 9: number analyzed (Participants) | 30 | 28
  My first treatment improved my appearance at Week 9 | 96.7 | 89.3
  I am satisfied with the contour of my lower face after treatment at Week 3 | 96.8 | 79.3
  I am satisfied with the contour of my lower face after treatment at Week 6: number analyzed (Participants) | 30 | 29
  I am satisfied with the contour of my lower face after treatment at Week 6 | 96.7 | 93.1
  I am satisfied with the contour of my lower face after treatment at Week 9: number analyzed (Participants) | 30 | 28
  I am satisfied with the contour of my lower face after treatment at Week 9 | 100 | 96.4
  I am satisfied with how well-defined my chin looks at Week 3 | 93.5 | 37.9
  I am satisfied with how well-defined my chin looks at Week 6: number analyzed (Participants) | 30 | 29
  I am satisfied with how well-defined my chin looks at Week 6 | 93.3 | 86.2
  I am satisfied with how well-defined my chin looks at Week 9: number analyzed (Participants) | 30 | 28
  I am satisfied with how well-defined my chin looks at Week 9 | 96.7 | 89.3
  I feel more attractive after treatment at Week 3 | 80.6 | 72.4
  I feel more attractive after treatment at Week 6: number analyzed (Participants) | 30 | 29
  I feel more attractive after treatment at Week 6 | 93.3 | 75.9
  I feel more attractive after treatment at Week 9: number analyzed (Participants) | 30 | 28
  I feel more attractive after treatment at Week 9 | 90.0 | 85.7
  I feel comfortable being photographed at Week 3 | 77.4 | 55.2
  I feel comfortable being photographed at Week 6: number analyzed (Participants) | 30 | 29
  I feel comfortable being photographed at Week 6 | 86.7 | 75.9
  I feel comfortable being photographed at Week 9: number analyzed (Participants) | 30 | 28
  I feel comfortable being photographed at Week 9 | 90.0 | 78.6
  Compared to my first treatment, treating both areas in combination improved my appearance at Week 6: number analyzed (Participants) | 30 | 29
  Compared to my first treatment, treating both areas in combination improved my appearance at Week 6 | 100.0 | 89.7
  Compared to my first treatment, treating both areas in combination improved my appearance at Week 9: number analyzed (Participants) | 30 | 28
  Compared to my first treatment, treating both areas in combination improved my appearance at Week 9 | 100.0 | 92.9
  I am satisfied with the shape of my chin at Week 3 | 96.8 | 41.4
  I am satisfied with the shape of my chin at Week 6: number analyzed (Participants) | 30 | 29
  I am satisfied with the shape of my chin at Week 6 | 96.7 | 89.7
  I am satisfied with the shape of my chin at Week 9: number analyzed (Participants) | 30 | 28
  I am satisfied with the shape of my chin at Week 9 | 100.0 | 92.9

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to Week 9
Description: Safety population was defined as all participants who were injected with study product.
Arm/Group | Down-up | Top-down
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 7/32 | 5/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Down-up (N=32) | Top-down (N=29)
Implant site bruising (General disorders) | 1 (1) | 2 (2)
Implant Site Pain (General disorders) | 6 (6) | 3 (3)
Implant site swelling (General disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT04520997/Prot_SAP_001.pdf